CLINICAL TRIAL: NCT06107101
Title: Investigating the Effects of Th2 Modulation on the Generation and Persistence of Tissue Adaptive Immune Memory in Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: th2 Modulation CRSwNP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Paul's Sinus Centre (Other)
Responsible Party: Principal Investigator, Dr. Andrew Thamboo, MD, Clinical Assistant Professor, St. Paul's Sinus Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H23-01777
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: * Treatment group:20 subjects with CRSwNP and asthma that will start Mepolizumab treatment
  * Disease control group: 10 subjects with CRSsNP without asthma that will not start Mepolizumab and will continue their standard of care treatment.
  * Control group: 10 healthy subjects without any sinus disease
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment (Experimental): 20 subjects with CRSwNP and asthma that will start Mepolizumab treatment
  Interventions: Drug: Mepolizumab
- Disease control group (No Intervention): 10 subjects with CRSsNP without asthma that will not start Mepolizumab and will continue their standard of care treatment.
- Control group (No Intervention): 10 healthy subjects without any sinuses disease

INTERVENTIONS:
Drug: Mepolizumab — 100mg of mepolizumab every 4 weeks subcutaneously for 6 months
  Arms: Treatment

SUMMARY:
Chronic rhinosinusitis (CRS) is a condition of persistent sinonasal mucosal inflammation which affects 11.9% of the US population. Mepolizumab is newly approved to treat chronic rhinosinusitis with nasal polyps (CRSwNP, the spaces inside nose and head are swollen and inflamed) and acts booking interleukin-5 (IL-5) a protein implicated in the inflammatory process. We aim to use Single-cell RNA sequencing (RNA-Seq, a method of genetically 'barcoding' cells to allow gene expression to be profiled at the level of individual cells) to study the effects of IL-5 blockade on the generation and maintenance of nasal adaptive immune responses, in CRS subjects.

DETAILED DESCRIPTION:
Purpose:

CRS is a poorly understood disease with suboptimal therapeutic strategies and a high disease burden. Adaptive immunity in the form of Th2 polarized T cell responses and B cell IgE class switching, and plasma cell infiltration, are a core component of eosinophilic CRS and asthma, yet our understanding of adaptive immunity in CRS remains limited. Modulating the Th2 response, through IL-5 blockade, leads to mixed results for CRSwNP patients. There are a number of patients who achieve improved asthma control with IL-5 blockade therapies that fail to see the same improvements in their nasal disease, outlining the currently limited understanding of factors involved in disease activity, disease endotypes, and the effects of modulating the Th2 response in this tissue environment. Improved understanding of nasal tissue immunity modulation by IL-5 blockade at a cellular level is an essential step towards appropriate patient selection and development of new targeted therapeutics. Single-cell transcriptomics is powerful tool for characterizing tissue immune landscapes and functional variations, has as yet been poorly utilized beyond studies of nasal epithelium in CRS

Hypothesis

* IL-5 blockade stimulates increased activity of nasal tissue T cells > peripheral blood T cells, and promotes increased tissue T cell Th2 polarization
* IL-5 blockade stimulates increased B cell germinal center activity in nasal secondary and tertiary lymphoid structures, through increased Tfh-B cell interactions and increased maturation to tissue antibody-secreting cells through BLIMP1 upregulation in Germinal Centre B cells.

Objectives

1. Characterise the local mucosal B cell response in tertiary (nasal) and secondary (postnasal space) lymphoid organs in CRSwNP, compared with circulating immunity, through visualization and modeling of germinal center activity, cellular support for germinal center activity and assessment of B cell clonal selection, class-switching, fate, and somatic hypermutation using single-cell transcriptomics, single-cell BCR (B- cell receptor) sequencing and spatial resolution through confocal microscopy.
2. Use single-cell transcriptomics and VDJ (variable, diversity, and joining) repertoire analysis to characterize the effects of Th2 modulation, through IL-5 blockade, on the formation and maintenance of nasal T and B cell adaptive immune memory.
3. Localize nasal sources of pro-inflammatory signaling in CRSwNP in the presence of IL-5 blockade, using single-cell transcriptomics, confocal microscopy, and nasal cytokine analysis.
4. Compare nasal pro-inflammatory cell subsets with paired peripheral blood samples by single cell transcriptomics, to correlate activity with biomarker candidates.

Research design

The proposed study is a prospective experimental medicine study using IL-5 blockade as a way of investigating the effects of Th2 modulation on the generation of local tissue adaptive immunity in CRSwNP. Participants will be classified in:

* Treatment group:20 subjects with CRSwNP and asthma that will start Mepolizumab treatment
* Disease control group: 10 subjects with CRSsNP without asthma that will not start Mepolizumab and will continue their standard of care treatment.
* Control group: 10 healthy subjects without any sinuses disease

This study involves three study visits for the Treatment arm (Baseline, weeks 6, and 30), two visits for disease control subjects, and one (Baseline) visit for Healthy control subjects.

Participants on study medication will receive 100mg of mepolizumab every 4 weeks subcutaneously.

Treatment Arm:

CRSwNP (NPS 1-8) and asthma undergoing IL-5 blockade (Mepolizumab)

• Week 0: Recruitment, screening, and initiating standard-of-care therapy

o Nasal and blood samples Week 6 - Pre-Mepolizumab commencement (Pre-treatment) Week 30 - After Mepolizumab commencement (On treatment)

Control Arm:

1. Diseased Control:

   CRSsNP without asthma

   • Week 0: Recruitment, screening, and initiating standard-of care therapy

   o Nasal and blood samples Week 6 - After 6 weeks standard of care therapy
2. Healthy control • Week 0: Recruitment and screening, Nasal and blood samples

Statistical analysis Single cell RNA sequencing data Sequenced data will be aligned with CellRanger v7.0. The resulting output files will be processed using a standard filtering and QC pipeline in Scanpy. The batch correction will be performed using scVI, and Leiden clustering will be performed. Cluster labels will be assigned using canonical marker genes and published gene signatures, with validation using a published dataset of sorted immune cells via the SingleR package. The downstream analysis will include, but not be limited to, gene set expression analysis (GSEA) of Hallmark and Gene Ontology genesets, differential abundance testing, weighted gene co-expression network analysis, and imputation of cell-cell interaction using CellphoneDB. TCR analysis will be performed using Scirpy, and BCR analysis with the Dandelion, and Immcantation suites

ELIGIBILITY:
Inclusion Criteria:

* Participants must be >=19 of age at the time of signing the informed consent form.
* Capable of giving signed informed consent.
* Treatment group:

  1. Bilateral Chronic Rhinosinusitis with Nasal Polyposis and Asthma

     a. Diagnosis consistent with EPOS 2020 b. Endoscopic Nasal Polyps Score (1-8) c. Asthma diagnosis based on: i. Consistent Clinical symptoms (History of wheeze, cough and breathlessness) ii. Reversible airflow obstruction (Spirometry)
  2. Eligibility for Mepolizumab therapy (Canada)
  3. On waiting list for surgery with planned wait of >6 months
* Disease control group:

  * Bilateral Chronic Rhinosinusitis without Nasal Polyposis, (only for the disease control group) oDiagnosis consistent with EPOS 2020

Healthy controls:

* Participants >=19 of age and capable of giving signed informed consent
* Participants with no history of sinonasal or lower airway disease

Exclusion Criteria:

* Participants are excluded from the trial if any of the following criteria apply:

  1. Women who are pregnant, plan to become pregnant or breastfeed during the trial.
  2. Current participation in any other interventional treatment trials.
  3. Compliance: is unlikely to comply with trial visits based on investigator judgment.
  4. Secondary, or suspected secondary, cause of nasal polyposis:

     1. EGPA, positive MPO ANCA or circulating eosinophilia >10% total leukocytes
     2. Known or suspected hereditary ciliary dysmotility (e.g: Cystic fibrosis, childhood-onset nasal polyposis)
     3. Diagnosed or suspected malignant or premalignant nasal disease (e.g: Schniderian Papilloma, unilateral nasal polyposis)
     4. Fungal rhinosinusitis (CT/Histology), positive Aspergillus skin prick testing and/or positive Aspergillus IgE RAST testing.
     5. Aspirin Exacerbated Respiratory Disease/Salicylate allergy
  5. Known hypersensitivity or significant allergies to monoclonal antibodies.
  6. Malignant neoplasm within 5 years (from screening) excluding basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterine cervix treated locally and without metastatic disease for 3 years.
  7. A history of a primary immunodeficiency.
  8. Active bleeding disorders, and/or inability to support interruption to anticoagulant or anti-platelet therapies for nasal biopsy.
  9. Severe nasal deformity precluding endoscopic assessment/biopsy of postnasal space
  10. Severe heart failure (New York Heart Association Class IV) or other severe, uncontrolled cardiac disease.
  11. Have a history of a major organ transplant or hematopoietic stem cell/marrow transplant.
  12. Have an acute or chronic infection (excluding that related to CRS) requiring management as follows:

      * Currently on any treatment for a chronic infection such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria
      * Hospitalisation solely for treatment of proven infection requiring parenteral (IV or IM) antibiotics (antibacterial, antiviral, antifungal, or anti-parasitic agents) within 60 days of Day 1.
      * Proven severe infection requiring outpatient treatment with parenteral (IV or IM) antibiotics (antibacterial, antiviral, antifungal, or anti-parasitic agents) within 60 days of Day 1. Prophylactic anti-infective treatment is allowed.
  13. Known positive human immunodeficiency virus (HIV) status.
  14. Known positive Hepatitis B (HB) or Hepatitis C status.
  15. Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not related to asthma which, in the opinion of the principal investigator, could confound the results of the trial or put the participant at undue risk.
  16. Have a planned surgical procedure, laboratory abnormality, or condition that, in the opinion of the principal investigator, makes the participant unsuitable for the trial.
  17. Have received any monoclonal antibody therapy ever.
  18. Have received any investigational agent (that is not approved for sale in Canada) within 60 days of Day 1.
  19. Have previously undergone sinus surgery or nasal polypectomy
  20. Previous immunomodulatory therapy (excluding corticosteroids)

Healthy controls exclusion criteria

1. Have previously undergone sinus surgery or nasal polypectomy
2. Have received any monoclonal antibody therapy (e.g., dupilumab, mepolizumab, omalizumab)
3. Have known hypersensitivity or significant allergies to monoclonal antibodies
4. Have a positive human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C status
5. Have tumors in the nasal cavity
6. Participants currently participating in other clinical trials
7. Have severe, uncontrolled cardiac disease
8. Have a history of a major organ transplant or hematopoietic stem cell/marrow transplant
9. Have an acute or chronic infection that is not related to chronic rhinosinusitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Endotyping nasal response to Mepolizumab | week 30
  Clinical response vs standard of care change in Endoscopic Nasal Polyp Score
Endotyping nasal response to Mepolizumab | week 30
  Clinical response vs standard of care change in SNOT-22 score
Endotyping nasal response to Mepolizumab | week 30
  Clinical response vs standard of care change in degree os eosinophil depletion
Nasal immune endotyping | week 30
  Comparison of Circulating B cells, Pre-IL-5 subjects, CRSsNP subjects, Healthy controls, Nasal vs NALT

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Sinus Centre, Vancouver, British Columbia, Canada